CLINICAL TRIAL: NCT04622787
Title: Implementation of Early Detection and Early Intervention Service Delivery in Infants at Risk for Cerebral Palsy to Promote Infants' Psychomotor Development and Maternal Health
Acronym: BornTogether
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Pisa (Other)
Collaborators: European Commission (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Andrea Guzzetta, Associate Professor, University of Pisa
Other Study IDs: BornTogether; 848201 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2020-07-30; First posted 2020-11-10 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Tuscany, Italy: Infants at risk of Cerebral Palsy in Tuscany, Italy
- Infants at risk of Cerebral Palsy in Georgia: Infants at risk of Cerebral Palsy in Georgia
- Sri-Lanka: Infants at risk of Cerebral Palsy in Sri-Lanka
- Denmark: Infants at risk of Cerebral Palsy in Denmark
- Infants at risk of Cerebral Palsy in the Netherlands: the Netherlands
- remote Queensland, Australia: Infants at risk of Cerebral Palsy in remote Queensland, Australia
- Medical professionals: Medical/healthcare providers from all involved geographic locations that work with infants at risk or with diagnosis of cerebral palsy will be provided opportunities for the participation in face-to-face and/or e-learning platform trainings on the the international early detection guidelines.
  Interventions: Other: Knowledge translation

INTERVENTIONS:
Other: Knowledge translation — A. Healthcare Providers Observational Study - measure of the effectiveness of the International Guidelines training courses (face to face and online) delivered to medical professionals (involves all clinical partners).
  The International Guidelines training courses on the evidence-based principles of Early Detection (ED), Early surveillance (ES), and Early intervention (EI) will be delivered to healthcare providers.
  Face-to-face professional trainings will be set up at each Consortium partner location. E-learning platform will allow for training and follow-up resources will be available to clinicians in all languages that are spoken/written in the locations of the Consortium partners.
  Clinicians will be assessed on their knowledge and standard clinical practices in survey format before trainings and after the trainings.
  Groups: Medical professionals

SUMMARY:
The BORNTOGETTHERE consists of improving health programs for early detection and surveillance of Cerebral Palsy (CP) by implementing the first International Clinical Practice Guidelines (Novak et al, 2017) in multiple sites in Europe (Italy, Denmark, Netherlands), in low- and middle-income countries (Georgia, Sri Lanka) and hard to reach populations (Remote Queensland, QLD and Western Australia, WA). In addition, exploiting early detection of infants at very high risk of CP, the investigators will implement best-evidence knowledge on early intervention in CP, thereby improving the outcomes of the infants and of their caregivers.

DETAILED DESCRIPTION:
The overall aim of the study is to utilize Knowledge Translation strategies to disseminate culturally appropriate guidelines for early detection, surveillance, and early intervention for infants at risk for CP.

Primary objectives A1 To optimize the context-specific health programs for early detection of CP through the implementation of a tailored multifaceted knowledge translation strategy, in >500 infants with CP from Tuscany (Italy); Denmark; Netherlands, Georgia, Sri Lanka, and rural/ remote Australia (QLD, WA).

The investigators will also evaluate health care resource usage following the implementation of our translation strategy compared with a two-year period prior to the implementation- e.g. costs of early detection and targeted surveillance, targeting infants with CP (costs and consequences/outcomes of surveillance and intervention).

H1 Our hypothesis is that, compared with usual care, implementation of our translation strategy will increase the proportion of children that receive a diagnosis of CP <6 months of age from ~25% to >60%, as measured by CP Registers. Additional costs of screening and surveillance in our translation strategy will be off-set by targeting the highest risk babies earlier. Health care costs and usage will be focused on the most at-risk group, leading to improved outcomes across all children (costs/consequences analysis).

A2 To optimize the context-specific health programs for early surveillance of associated impairments and functional limitations of infants with CP, thereby fostering individualised (needs-based patient specific) early intervention and preventing secondary complications (e.g. hip dislocation, feeding disorders). The investigators will evaluate the early developmental trajectory of CP in infants aged 0-2 years and parental mental health to inform early intervention and surveillance needs to improve prediction of outcomes. The investigators will also compare the rates of hip displacement at 2 years following the implementation of our translation strategy compared with usual care (i.e. proportion of children with migration percentage >30%).

H2 Our hypothesis is that the natural history of CP in infants aged 0-2 years will differ according to motor severity, with different trajectories identified as early as 6 months' corrected age. The investigators also predict a reduction in the rate of hip displacement from 33% in current practice to <10% following the implementation of our translation strategy (consistent with Scandinavian screening programs).

A3 To optimize the context-specific health programs for early intervention in infants with CP, thereby improving the outcomes of both the infant and the caregivers. In Low- and Middle-Income Countries (LMIC) and hard-to-reach populations the investigators will also implement a community-based, parent delivered early intervention program for infants at high risk of CP (LEAP-CP).

H3 Our hypothesis is that infants with CP who receive the multi-domain intervention will have better motor development (Peabody DMS), social- emotional development on the Infant-Toddler Social Emotional Assessment (ITSEA), cognitive development (Bayley Scale of Infant Development (BSID III)) compared to infants receiving care as usual. Caregivers who receive the multi-domain intervention will have reduced scores on the Depression, Anxiety and Stress Scale compared to caregivers receiving care as usual.

Based on the aims listed above, there will be 3 parallel studies within the protocol:

A: Healthcare Providers Observational Study B: Infant Prospective Observational study C: Infant wait-list Randomised Controlled Trial of LEAP-CP, a home - based early intervention (Georgia, Sri-Lanka and remote Australia only, RCT (randomized controlled trial) registered separately with ANZCTR)

ELIGIBILITY:
Healthcare providers Knowledge Translation:

Inclusion Criteria:

* Medical/healthcare provider or advanced trainee
* Works with infants at risk or with diagnosis of cerebral palsy
* Practices in Georgia, Sri-Lanka, The Netherlands, Denmark, Remote Queensland region of Australia, Tuscan region of Italy,

Exclusion Criteria:

* Not a healthcare provider or trainee
* Located (practicing) outside of study country locations

Infant and family observational study:

Inclusion criteria: Infants aged <12 months' corrected age at with one of the following

* Extremely preterm
* Extremely low birthweight
* Neonatal encephalopathy
* Stroke
* Abnormal General Movements with abnormal brain neuroimaging
* Abnormal General Movements with abnormal Neurological Evaluation
* Abnormal brain neuroimaging with abnormal Neurological Evaluation

Exclusion criteria

* Lethal abnormalities
* congenital conditions not associated with cerebral palsy (e.g. Down's Syndrome)
* complex medical conditions requiring acute medical care

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare providers Knowledge Translation: Medical/healthcare providers that work with infants at risk or with diagnosis of cerebral palsy in involved countries
  Infant and family observational study: Infants aged <12 months' corrected age until 24 months of age.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge Translation effectiveness | through study completion, an average of 3 years
  Clinicians will be tested in survey format on their knowledge of the guidelines

SECONDARY OUTCOMES:
Infant age at diagnosis of Cerebral Palsy | through study completion, an average of 3 years
  change in average age at CP diagnosis at location before clinicians' trainings and up to 2 years after clinicians' trainings

CONTACTS AND LOCATIONS:
Locations (1):
- Universitá di Pisa, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No
The Coordinator (and data controller) of BORNTOGEtTHERe will not collect personal data from the Consortium Partners. Personal data will be collected within each participating institution and stored locally according to Pseudonymized data will be provided from the participating partner institutions to the data controller (The Coordinator) for the BORNTOGEtTHERe project.

REFERENCES:
- See also: The General Data Protection Regulation (GDPR) — https://gdpr.eu